CLINICAL TRIAL: NCT03489278
Title: Clinical Procedures to Support Research in ALS (CAPTURE-ALS)
Brief Title: Clinical Procedures to Support Research in ALS
Acronym: CAPTURE-ALS
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Muscular Dystrophy Association (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Michael Benatar, Chief, Neuromuscular Division, University of Miami
Other Study IDs: 20170785; U54NS092091 (NIH)
Record Dates: First submitted 2018-03-23; First posted 2018-04-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS-Frontotemporal Dementia; Primary Lateral Sclerosis; Progressive Muscular Atrophy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional: Provide blood for a DNA sample during a clinic visit. Participants can choose to allow collection of information from their medical record, but choose not to give a blood sample for testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected: Affected with ALS or a related disorder.

SUMMARY:
The purpose of the Clinical Procedures To Support Research (CAPTURE) study is to utilize information collected in the medical record to learn more about a disease called amyotrophic lateral sclerosis (ALS) and related disorders.

DETAILED DESCRIPTION:
The study will consent patients with ALS or related disorders that are receiving care at a clinical center in the CReATe consortium that uses Epic as its electronic health record (EHR) system. The study aims to systematically gather a clinical dataset through the EHR using a standardized approach to characterize the natural history of ALS and related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS or a related disorder (e.g. primary lateral sclerosis, progressive muscular atrophy).
* Receiving care at a clinical center that uses Epic as its EHR.
* Able and willing to provide informed consent (or informed consent obtainable from a designated proxy).

Exclusion Criteria:

* Inability to understand English and/or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Affected patients receiving care at a clinical center that uses Epic as EHR.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Using the ALS Toolkit for collecting and using electronic health record data for research purposes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, MBChB, MS, DPhil, Principal Investigator — University of Miami
Locations (11):
- United States (11):
  - University of California, Irvine, Irvine, California
  - Stanford University, Palo Alto, California
  - California Pacific Medical Center, San Francisco, California
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Providence Health & Services, Portland, Oregon
  - University of Texas San Antonio Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No